CLINICAL TRIAL: NCT03792282
Title: Effectiveness of Time-Restricted Feeding(TRF) on Overweight/Obese Women with Polycystic Ovarian Syndrome(PCOS): a Randomized Controlled Trial
Brief Title: Time-Restricted Feeding(TRF) on Overweight/Obese Women with Polycystic Ovarian Syndrome (PCOS)
Acronym: TRF-PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYH2018-017
Record Dates: First submitted 2018-12-30; First posted 2019-01-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Overweight and Obesity
Keywords: Polycystic Ovary Syndrome; Overweight and Obesity; Time-Restricted Feeding; Intermittent fasting regimens
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity; Intermittent Fasting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRF (Experimental): Participants in this group will focus on time restricted feeding (TRF) in addition to daily calorie restriction.
  Interventions: Behavioral: Time Restricted Feeding
- Usual care (Active Comparator): Participants in this group will receive a general lifestyle counseling.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Time Restricted Feeding — Participants will receive a diet of 1200-1500kcal/d and be instructed to eat only during a window of 8 hours (Finishing the last meal before 4pm).
  Arms: TRF
Behavioral: Usual care — Participants receive a general lifestyle counseling.
  Arms: Usual care

SUMMARY:
The aims of the present study is to examine whether Time-Restricted Feeding (TRF) is a safe and effective regimen to improve insulin resistance and decrease body weight in overweight/obese Polycystic ovary syndrome (PCOS) patients over 16 weeks compared to reduced energy restriction.

DETAILED DESCRIPTION:
Intermittent fasting regimens involve periods fasting followed by periods of eating freely. Time-Restricted Feeding (TRF) is a new form of intermittent fasting and involves shortening the eating window to 4-10 h/day. TRF is a safe lifestyle intervention for weight loss in adults with obesity. Accumulating evidence suggests that TRF is an effective means of decreasing body weight and improving insulin resistance but did not have any negative impact on eating disorder symptoms, body image perception, or eating behaviors. Polycystic ovary syndrome (PCOS) is the most common endocrine condition in productive-aged women. About 60-70 % of women with PCOS are obese or overweight, and obesity is associated with insulin resistance. Since many women with PCOS seem to have insulin resistance, compensatory hyperinsulinemia is thought to contribute to hyperandrogenism by direct stimulation of ovarian production of androgens and by inhibition of liver synthesis of SHGB. It is important to ameliorate insulin resistance in PCOS patients.The aims of the present study is to examine whether TRF is a safe and effective regimen to improve insulin resistance and decrease body weight in overweight/obese PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI≥24kg/m2
* Polycystic ovary syndrome has been diagnosed

Exclusion Criteria:

* Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
* The body weight fluctuated more than 5% in recent 3 months.
* Liver and kidney dysfunction: renal impairment, creatinine clearance rate < 30 mL/min/1.73 m2, transaminase increased, more than three times higher than the normal limit;
* History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
* History of thyroid diseases;
* Having been in pregnancy.
* Researchers believe that there are any factors that affect assessing subjects' participation in trial.
* History of malignant tumors;
* History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
* Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight)
* Patients who cannot be followed for 16 months (due to a health situation or migration)
* Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women have the PCOS.
Enrollment: 93 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in body weight (Kilograms) | Baseline and 16 weeks
  Changes in body weight (Kilograms)
Change in insulin resistance | Baseline and 16 weeks
  Insulin resistance will be assessed by HOMA-IR

SECONDARY OUTCOMES:
Change in BMI | Baseline and 16 weeks
Changes in waist circumference (cm) | Baseline and 16 weeks
Changes in Waist-to-Hip Ratio(WHR) | Baseline and 16 weeks
Changes in systolic pressure（SBP） | Baseline and 16 weeks
Changes in diastolic pressure (DBP） | Baseline and 16 weeks
Change in Body fat percent | Baseline and 16 weeks
Change in Fat mass | Baseline and 16 weeks
Change in Skeletal muscle mass | Baseline and 16 weeks
Change in CHO level | Baseline and 16 weeks
Change in TG level | Baseline and 16 weeks
Change in HDL level | Baseline and 16 weeks
Change in LDL-c level | Baseline and 16 weeks
Change in Fasting Blood Glucose (FBG) level | Baseline and 16 weeks
Change in ALT level | Baseline and 16 weeks
Change in AST level | Baseline and 16 weeks
Change in GGT level | Baseline and 16 weeks
Change in Testosterone level | Baseline and 16 weeks
Change in Sex hormone binding globulin (SHBG) level | baseline and 16 weeks
Change in Free androgen index （FAI） | Basline and 16 weeks
Change in Ferriman-Gallway score （F-G score:） | Baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Changqin Liu, MD, Principal Investigator — The first afilliated hospital of Xiamen university
Locations (1):
- The first afilliated hospital of Xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717